CLINICAL TRIAL: NCT07004621
Title: Videolaryngoscopy Versus Direct Laryngoscopy for Endotracheal Intubation of Obese Patients: a Prospective Randomized Trial
Acronym: VL or DL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Skladzien, MD PhD, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1072.6120.135.2023 (Cracow)
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Intubating Laryngeal Airway
Keywords: laryngoscopy; tracheal intubation; o besity patients ,; v ideolaryngoscopes

STUDY DESIGN:
Intervention Model Description: The study group will be male and female patients, ASA II or III, over 18 years of age and under 75 years of age. Each patient will undergo abdominal (bariatric) surgery.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator): traditional laryngoscope for the first laryngoscopy
  Interventions: Other: measurment of intubation time in seconds
- Video-Laryngoscope (Experimental): video laryngoscope will be used to intubate half of the people
  Interventions: Other: measurment of intubation time in seconds

INTERVENTIONS:
Other: measurment of intubation time in seconds — determine whether modern technologies such as videolaryngoscopy shorten intubation time.

SUMMARY:
Patients were randomly assigned (1:1) to either a Macintosh laryngoscope group ("Macintosh group") or a videolaryngoscope group ("Video group").

DETAILED DESCRIPTION:
In the Macintosh group, intubation was performed with a standard curved Macintosh blade. In the Video group, intubation was performed with the assigned videolaryngoscope. If intubation proved difficult with the initially assigned device, anaesthesiologists could switch to the alternative method at their discretion (rescue technique).

ELIGIBILITY:
• Inclusion criteria: Adult patients (> 18 years) of both sexes with BMI > 35 kg/m² scheduled for laparoscopic sleeve gastrectomy (ASA < IV).

• Exclusion criteria:

* Patient's refusal to participate.
* Known allergy to drugs used during anaesthesia.
* Chronic pain syndromes.
* Chronic opioid use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
determine whether modern technologies such as videolaryngoscopy shorten intubation time. | 1 day
  measurment of intubation time in seconds

SECONDARY OUTCOMES:
complications | 1 day
  included the incidence of failed intubation with the assigned device, the number of intubation attempts, and the use of an introducer (bougie). Any intubation attempt that failed could be rescued with the alternative device.

CONTACTS AND LOCATIONS:
Locations (1):
- SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
Participatned did not agree

REFERENCES:
- [Background] Yumul R, Elvir-Lazo OL, White PF, Sloninsky A, Kaplan M, Kariger R, Naruse R, Parker N, Pham C, Zhang X, Wender RH. Comparison of three video laryngoscopy devices to direct laryngoscopy for intubating obese patients: a randomized controlled trial. J Clin Anesth. 2016 Jun;31:71-7. doi: 10.1016/j.jclinane.2015.12.042. Epub 2016 Mar 23. PMID 27185681